CLINICAL TRIAL: NCT05571891
Title: Effect of Intermittent Fasting (Month of Ramadan) on Health
Acronym: RAMA1
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Piero Portincasa, MD, PhD, Dr honoris.Causa., AGAF Professor of Internal Medicine Chief, Clinica Medica "A. Murri" Director, Dept. Biomedical Sciences & Human Oncology, University of Bari
Other Study IDs: RAMA-1 2022
Record Dates: First submitted 2022-09-15; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Fasting, Intermittent
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample collected for metabolic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, many studies have shown the positive effect of certain types of fasting on human health, particularly on obesity, diabetes, and aging. In particular, the beneficial effects of intermittent fasting are gaining more attention among clinical researchers. Intermittent fasting is the voluntary abstinence of individuals, from food (some or all food, drinks, or both) for a period longer than a typical overnight 12 h fast. The digestibility of food is an important characteristic, associated with the concepts of health and well-being. Digestive motility disorder leads to various digestive problems like difficulty in swallowing, acid reflux disease, severe constipation, diarrhea, abdominal pain, vomiting, and bloating. Hence the investigators aimed to assess the impact of intermittent fasting (religious fasting "Ramadan") on digestibility (gastrointestinal motility), weight, blood glucose level, gut microbiota, and gut permeability of the subjects. A cohort of 21 subjects homogeneously distributed by sex, age, and BMI will be prospectively enrolled and involved in the study. By comparing the analytical data before and after Ramadan the effect of intermittent fasting on digestibility, blood glucose and microbiota will be characterized by the investigators.

DETAILED DESCRIPTION:
The study has been developed as a clinical trial. It is expected the signing of the informed consent and authorization to the personal data (attached information form - Consent and information GDRP). A total of 21 subjects aged between 20 and 60 years homogeneous for sex (10M:11F) and body mass index (BMI = kg/m2) will be enrolled for the study. Subjects will be required to practice a 29/30 day religious fast.

All subjects will provide two stool samples for 16S rRNA sequencing, first at baseline and the second after 30 days of Ramadan for gut microbiota assessment. In addition, at the beginning of the study, subjects will be submitted to complementary and validated semi-quantitative questionnaires to assess the severity, frequency, and duration of the gastrointestinal symptoms in the month prior to the start of the study, the study of gastric and cholecystic motility, the assessment of the oro-cecal transit time. In addition, at the beginning of the study, during and after fasting, subjects will be complementary and validated semi-quantitative food questionnaires to evaluate the diet.

Gastric and cholecystic motility will be assessed using a portable ultrasound scanner (Esaote AU450 and Noblus, Hitachi Medical, Tokyo, Japan) equipped with a 3.5 MHz convex probe in order to measure time-dependent changes in fasting and post-meal cholecyst volumes and gastric antral areas. All experiments will begin at 08:00 after an overnight fast of 12 hours. Gastric and cholecyst motility will be compared after the standard meal (Nturi ENSUR) ingested along with a 120 ml glass of water in which 15 ml of lactulose will be dissolved. Lactulose provides a non-absorbable but fermentable substrate useful for measuring the oro-cecal transit time (OCTT). The solution will be drunk at room temperature for one minute in the presence of the examiner.

Transit times will be measured using breath testing, following standard guidelines. During the 30 days prior to the test, subjects should not take antibiotics, probiotics, prokinetics, or other medications that affect gastrointestinal motility and gut microbiota. To avoid prolonged intestinal production of H2 due to the presence of non-absorbable or slowly fermentable foods, each subject should follow a special diet the day before the test consisting of meat, fish, and olive oil. No other fermentable foods or sugary drinks will be allowed. Breath samples will be taken before ingestion of the test meal and then every 15 minutes for 120 minutes after ingestion of the meal using a pre-calibrated portable hydrogen-sensitive electrochemical device (EC60-Gastrolyzer, Bedfont, USA). Results will be expressed as excretion of H2 in parts per million (p.p.m). The 10 p.p.m increase from baseline over two consecutive measurements will provide the OCTT for each subject after conversion to minutes.

In order to evaluate the impact of Ramadan, parameters related to glycemia, triglycerides, and cholesterol will be evaluated by a blood test. Fecal microbiota analysis will be conducted at DISSPA (Department of Soil, Plant, and Food Sciences).

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to provide informed consent
* Age between 20 and 60
* Healthy Volunteers

Exclusion Criteria:

* Lack of informed consent
* Diagnosis of organic diseases, including neoplastic inflammatory diseases or cardiovascular diseases
* Medications that can affect the gastrointestinal tract and interfere with symptoms
* Pregnancy
* Presence of diseases with a prognosis of less than 12 months
* Celiac disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For this pilot study 21 subjects homogeneously distributed by sex, age and BMI will be involved. The subjects will be required to practice religious fasting (Ramadan fasting) for 29/30 days.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Effect of intermittent fasting on anthropometric measurements | 1 months
  height and weight will be combined to calculate Body Mass Index (BMI, expressed as Kg/m^2). measurements will be recorded in all subjects at enrollment and at the end of the intermittent fasting
Effect of intermittent fasting on gastric intestinal motility | 1 month
  The gastric and cholecystic motility was assessed by ultra sound scanner and the severity, frequency and duration of gastrointestinal symptoms was using the questionnaires before and after the intermittent fasting
Effect of intermittent fasting on gut microbiome | 1 month
  Analysis of the gut microbiome by DNA extraction from faecal samples and high-throughput rRNA gene-targeted amplicon sequencing Gut metabolome: Faecal samples will be analysed by GC-MS and 1H-NMR. Faecal SCFA will be also analysed.
Effect of intermittent fasting on visceral and subcutaneous fat quantity and deposition | 1 month
  The visceral fat (VAT) and subcutaneous fat (SAT) deposition on different parts of the body such as pre-hepatic, pre-pancriatic, pre-aortic, hepato-renal, and spleno-renal fats will be analysed by ultrasound ecography. The amount of SAT and VAT will be expressed in mm before and after intermittent fasting.
Effect of intermittent fasting on serum gluco-lipid profile | 1 month
  Serum glucose (mg/dL), total cholesterol (mg/dL), LDL cholesterol (mg/dL), HDL cholesterol (mg/dL), triglycerides (mg/dL) will be measured at enrollment and at the end of the intermittent fasting.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences and Human Oncology - Clinica medica "A. Murri", Bari, BA, Italy